CLINICAL TRIAL: NCT04874701
Title: Effects of Capsimax on Appetite, Energy Intake and Blood Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: OmniActive Health Technologies (Industry)
Responsible Party: Principal Investigator, Angelo Tremblay, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAPSIMAX
Record Dates: First submitted 2021-04-25; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Obesity; Body Weight; Weight Loss; Overweight
MeSH Terms: conditions — Obesity; Body Weight; Weight Loss; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capsimax (Experimental)
  Interventions: Drug: Capsimax; Other: Energy restriction
- Placebo (Placebo Comparator): Placebo, 2 capsules per day, for 12 weeks
  Interventions: Other: Energy restriction

INTERVENTIONS:
Drug: Capsimax — Capsimax, 2 capsules per day, for 12 weeks Medicinal ingredient: Capsicum annuum Quantity (per capsule): 100.0 mg
  Arms: Capsimax
Other: Energy restriction — Personalised diet plan targeting a 500 kcal/day energy restriction

SUMMARY:
Obesity is an ongoing major public health problem in most countries of the world for which the agrifood industry still remains criticized because of the abundant offer of high sugar-lipid-energy dense foods, particularly in the fast-food sector. The resulting societal pressure on the food industry probably explains in part the efforts that have been deployed to seek natural active ingredients and to develop functional foods favorably influencing energy balance. Capsaicin is a food non-nutrient constituent that was shown to decrease appetite sensations and subsequent energy intake. The measurement of heart rate variability revealed an association between the increase in sympathetic nervous system (SNS) activity and the satiating effects induced by capsaicin. This is concordant with the observation that pre-prandial intake of capsaicin, be it in capsules or diluted in tomato juice, increased satiety and reduced energy intake.

The objective of this study is to evaluate the long effects of Capsimax on appetite sensations and energy expenditure under conditions of moderate energy restriction and to evaluate the long-term effects of Capsimax on energy intake and expenditure under conditions of moderate energy restriction.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women
* Between 18 and 50 years
* Healthy
* Non-smoker
* BMI between 25 and 35 kg/m2
* Weight stability

Exclusion Criteria:

* Pregnant or menopausal woman
* History of losing and gaining weight (yo-yo)
* Taking medication for diabetes, hypertension, depression, or hypothyroid
* Taking a supplement for weight loss
* Vegetarian, vegan, intolerant to gluten or pepper (investigational product), and severe allergy to peanuts or nuts
* Suffers from Irritable Bowel Syndrome or gastro-oesophageal reflux
* Suffers from stomach ulcers or inflammation
* Other serious conditions such as cardiovascular, renal, liver, and lung diseases
* History of drug abuse and current alcohol abuse
* Use of any medication (including over-the-counter medications and herbal remedies) such as grapefruit juice, piperine, NSAIDs, etc.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2018-01-07 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in appetite sensations, energy intake and food preferences at Week 12 | 12 weeks
  Visual analog scales used after a standardized breakfast and a buffet-type meal to measure hunger, fullness, satiety and desire to eat.
Change from Baseline in energy expenditure at Week 12 | 12 weeks
  Energy expenditure measured at fasting stade, after a 15 minutes rest, by indirect calorimetry
Change from Baseline in Body weight and fat at Week 12 | 12 weeks
  Body weight and fat measured with Dual-energy X-ray absorptiometry (DXA)
Change from Baseline in Blood pressure at Week 12 | 12 weeks
  Blood pressure measured every 30 minutes during a 3h testing

SECONDARY OUTCOMES:
Change from Baseline Microbiota analysis at Week 12 | 12 weeks
  Sequencing of the 16S DNA to evaluate the evolution of the microbiota according to the diet.
Change from Baseline System analysis of endocannabinoids at Week 12 | 12 weeks
  The evaluation of the endocannabinoid system done on OpenArray TaqMan according to the expression in RNA of about fifty genes of this system and by their quantification by HPLC coupled to MS / MS mass spectrometry and / or by ion capture. IT-TOF
Change from Baseline sleeping quality (PSQI) at Week 12 | 12 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a validated questionnaire which evaluates sleep quality and disturbance over a 1-month time interval. The PSQI gives a score for seven different components : subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping.
  medication, and daytime dysfunction
Change from Baseline Feeding behaviors (TFEQ and Food cravings questionnaire) at Weeks 12 | 12 weeks
  Feeding behaviors measured by two validated questionnaires : The Three Factor Eating Questionnaire (TFEQ) which measures three main dimensions of human eating behaviors such as cognitive restraint, disinhibition and susceptibility for hunger and the Food cravings questionnaire
Change from Baseline anxiety (BDI and STAI) at Week 12 | 12 weeks
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. It can be used in clinical settings to diagnose anxiety and to distinguish it from depressive syndromes. The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Tremblay, Principal Investigator — Laval University
Locations (1):
- PEPS-Université Laval, Québec, Canada

IPD SHARING:
Plan to Share IPD: No